CLINICAL TRIAL: NCT05955404
Title: Effect of Kangaroo Mother Care in Alleviating Preterm Infant's Pain
Brief Title: Kangroo Mother Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hiba Abdulwahid Dawood, Principal Investigator, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: kangroo mother care
Record Dates: First submitted 2023-07-10; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Preterm Birth Complication
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: This study uses the Kangaroo mother care as a non-pharmacological strategy to alleviate the pain that preterm infants experience in the NICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kangaroo mother care (Experimental): This study uses the Kangaroo mother care as a non-pharmacological strategy to alleviate the pain that preterm infants experience in the NICU.
  Interventions: Other: Kangaroo mother care

INTERVENTIONS:
Other: Kangaroo mother care — This study uses the Kangaroo mother care as a non-pharmacological strategy to alleviate the pain that preterm infants experience in the NICU.

SUMMARY:
infants had a condition that might influence their responses to pain, e.g., congenital anomalies or severe illnesses requiring treatment with antiepileptics, muscle relaxants, or analgesic drugs.

DETAILED DESCRIPTION:
infants had a condition that might influence their responses to pain, e.g., congenital anomalies or severe illnesses requiring treatment with antiepileptics, muscle relaxants, or analgesic drugs and comparing the pain intensity with preterm infants who receive conventional care.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants whose corrected gestational age from (32 - <37) weeks of pregnancy
* Preterm infants who do not experience any painful procedure for last 24 hours
* Preterm infants do not receive any sedation for last 24 hours

Exclusion Criteria:

* full-term infants whose corrected gestational age is >37 weeks
* extremely preterm (< 28 weeks)
* very preterm (28-<32 weeks)
* proven or suspected sepsis
* major congenital malformations
* all heart defect except neonatal Patent ductus arteriosus (PDA)
* necrotizing enterocolitis
* neurodevelopmental disability
* who receive respiratory support {Mechanical Ventilation, Continuous Positive Airway Pressure, or high-flow support
* indicated for surgery
* contraindication to oral sucrose
* Twins
* infants had a condition that might influence their responses to pain, e.g., congenital anomalies or severe illnesses requiring treatment with antiepileptics, muscle relaxants, or analgesic drugs

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile-Revised (PIPP-R) | Two months
  The Premature Infant Pain Profile-Revised (PIPP-R) measures the intensity of pain that the preterm infants experience in NICU through infant indicators (change in heart rate from baseline, decrease in oxygen saturation from baseline, browse bulge, eye squeeze, and naso-labial furrow. It also includes gestational age and behavioral state.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing- The University of Baghdad, Baghdad, Iraq